CLINICAL TRIAL: NCT00045461
Title: A Randomized Phase II/III Trial Comparing Carboplatin-Ifosfamide (IC)-Chemotherapy Vs. IC-Chemotherapy Combined With Extreme Whole Body Hyperthermia In Patients With Recurrence Of Epithelial Ovarian Carcinoma: DOLPHIN-1-STUDY
Brief Title: Combination Chemotherapy With or Without Whole-Body Hyperthermia in Treating Patients With Recurrent Ovarian Epithelial, Fallopian Tube, or Peritoneal Cancer
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: LMU-DOLPHIN-1; CDR0000256532 (Registry Identifier: PDQ (Physician Data Query)); EU-20220
Record Dates: First submitted 2002-09-06; First posted 2003-01-27 (Estimated); Last update posted 2013-08-07 (Estimated); Status verified 2002-10

CONDITIONS: Fallopian Tube Cancer; Ovarian Cancer; Primary Peritoneal Cavity Cancer
Keywords: recurrent ovarian epithelial cancer; recurrent fallopian tube cancer; stage IIIA fallopian tube cancer; stage IIIB fallopian tube cancer; stage IIIC fallopian tube cancer; stage IV fallopian tube cancer; recurrent primary peritoneal cavity cancer; stage IIIA primary peritoneal cavity cancer; stage IIIB primary peritoneal cavity cancer; stage IIIC primary peritoneal cavity cancer; stage IV primary peritoneal cavity cancer; stage IIIA ovarian epithelial cancer; stage IIIB ovarian epithelial cancer; stage IIIC ovarian epithelial cancer; stage IV ovarian epithelial cancer
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — Carboplatin; Ifosfamide; Diathermy

INTERVENTIONS:
Drug: carboplatin
Drug: ifosfamide
Procedure: hyperthermia treatment

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Hyperthermia therapy kills tumor cells by heating them to several degrees above body temperature. Combining hyperthermia with chemotherapy may kill more tumor cells. It is not yet known if chemotherapy is more effective with or without whole-body hyperthermia therapy in treating gynecologic cancer.

PURPOSE: Randomized phase II/III trial to compare the effectiveness of chemotherapy with or without whole-body hyperthermia in treating patients who have recurrent ovarian epithelial, fallopian tube, or peritoneal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the time to progressive disease in patients with recurrent ovarian epithelial, fallopian tube, or extraovarian peritoneal cancer treated with carboplatin and ifosfamide with or without whole body hyperthermia.
* Compare the response rate, duration of response, and survival time of patients treated with these regimens.
* Compare the effect on the presence of disseminated tumor cells in bone marrow in patients treated with these regimens.
* Compare the toxicity of these regimens in these patients.
* Assess quality of life of patients treated with these regimens.

OUTLINE: This is a phase II safety and efficacy study followed by a phase III randomized, open-label, multicenter study.

* Phase II: Patients receive ifosfamide IV over 1 hour and carboplatin IV over 20 minutes on day 1. Patients also undergo whole body hyperthermia for at least 1 hour on day 1. Treatment repeats every 28 days for 6 courses in the absence of disease progression or unacceptable toxicity.
* Phase III (after successful treatment of 15 patients in phase II): Patients are stratified according to disease-free interval (6-12 months vs more than 12 months), measurable disease (bidimensionally measurable vs measurable by other clinical means), and disease recurrence (first recurrence vs second or greater recurrence). Patients are randomized to 1 of 2 treatment arms.

  * Arm I: Patients receive ifosfamide, carboplatin, and whole body hyperthermia as in phase II.
  * Arm II: Patients receive ifosfamide and carboplatin as in arm I.
  * In both arms, treatment repeats every 28 days for 6 courses in the absence of disease progression or unacceptable toxicity.

Quality of life is assessed before each course, 4 weeks after the last course, and then every 3 months for 2 years.

Patients are followed at 4 weeks and then every 3 months for 2 years.

PROJECTED ACCRUAL: A total of 15 patients will be accrued for phase II of this study. A total of 226 patients (113 per treatment arm) will be accrued for phase III of this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed ovarian epithelial, fallopian tube, or extraovarian peritoneal cancer

  * Recurrent disease (any FIGO stage)
  * Not amenable to curative surgery or radiotherapy alone
* Failed prior primary platinum-based therapy at least 6 months after therapy discontinuation
* Measurable lesion by CT scan, MRI, chest x-ray, or sonography

  * Physical examination allowed for documenting lymph node and skin metastases
  * Physical gynecological examination allowed for well-defined palpable tumor lesions
  * Increase in CA 125 without any measurable tumor is not acceptable as indication of recurrence
* No CNS metastases
* No tumor of borderline malignancy

PATIENT CHARACTERISTICS:

Age

* 18 to 65

Performance status

* ECOG 0-2

Life expectancy

* At least 24 weeks

Hematopoietic

* Neutrophil count at least 1,500/mm3
* Platelet count at least 100,000/mm3

Hepatic

* Not specified

Renal

* Creatinine clearance at least 60 mL/min
* No chronic or acute renal failure

Cardiovascular

* Cardiovascular function sufficient for hyperthermia treatment by stress-ECG
* No cardiomyopathy with impaired ventricular function
* No New York Heart Association class III or IV heart disease
* No cardiac arrhythmias influencing LVEF and requiring medication
* No myocardial infarction or angina pectoris within the past 6 months
* No uncontrolled arterial hypertension

Pulmonary

* Pulmonary function sufficient for hyperthermia treatment by pulmonary function tests

Other

* No untreated endocrinological disease (e.g., hyperthyroidism or diabetes mellitus)
* No other primary malignancy except carcinoma in situ of the cervix or adequately treated basal cell skin cancer
* No contraindication against hyperthermia treatment (e.g., photodermatosis, history of malignant hyperthermia, or claustrophobia)
* No hypersensitivity to carboplatin, ifosfamide, or any other study medication
* Not pregnant or nursing

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* See Disease Characteristics
* No concurrent cytotoxic or other antineoplastic therapy

Endocrine therapy

* Concurrent hormone replacement therapy allowed
* Concurrent steroid antiemetics allowed

Radiotherapy

* See Disease Characteristics
* At least 1 year since prior radiotherapy (tumoricidal dose) of the pelvis
* Concurrent palliative local radiotherapy for painful (nonprogressive) existing lesion is allowed if other measurable sites are present
* No concurrent radiotherapy to a second existing lesion

Surgery

* See Disease Characteristics

Other

* No prior form of hyperthermic therapy
* At least 3 weeks since other medications as part of another clinical study
* At least 3 weeks since prior investigational agents
* At least 6 weeks since prior betablockers
* No concurrent photosensitizing drugs
* No concurrent betablockers
* No other concurrent anticancer therapy

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 241 (Estimated)
Dates: Start 2000-06

PRIMARY OUTCOMES:
Time to progressive disease
Response rate
Duration of response
Survival time
Effects on the presence of disseminated tumor cells in bone marrow
Toxicity
Quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Harald Sommer, MD, Study Chair — Ludwig-Maximilians - University of Munich
Locations (7):
- Germany (5):
  - Charite University Hospital - Campus Virchow Klinikum, Berlin
  - Krankenhaus Nordwest, Frankfurt
  - University Medical Center Hamburg - Eppendorf, Hamburg
  - Universitaets - Kinderklinik - Luebeck, Lübeck
  - Kreiskrankenhaus Trostberg, Trostberg an der Alz
- Peterfy Korhaz Szulo-Nobeteg Oztaly, Budapest, Hungary
- Academisch Medisch Centrum at University of Amsterdam, Amsterdam, Netherlands